CLINICAL TRIAL: NCT01408641
Title: A 14-week Randomized, Placebo-controlled Study of Topiramate for Alcohol Use Disorders in Veterans With Posttraumatic Stress Disorder
Brief Title: Topiramate for Alcohol Use in Posttraumatic Stress Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator was deployed overseas
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, MPRC, Physician, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00047672
Record Dates: First submitted 2011-08-01; First posted 2011-08-03 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Dependence; Alcoholism; Alcohol Abuse; Alcohol Use Disorder; PTSD; Posttraumatic Stress Disorder
Keywords: topiramate; PTSD; drinking; alcohol
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental): Topiramate arm will be titrated (dose will increase slowly) over 6 weeks to 400mg or highest tolerated dose.
  Interventions: Drug: Topiramate
- Placebo (Sugar Pill) (Placebo Comparator): Placebo arm will receive matching capsules without topiramate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — Topiramate titrated over 6 weeks to 400mg or highest tolerated dose.
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo — Placebo capsules without topiramate
  Arms: Placebo (Sugar Pill)

SUMMARY:
Alcohol abuse and dependence (alcohol use disorders, AUDs) and posttraumatic stress disorder (PTSD) are both prevalent in Veterans. Treating AUDs in Veterans with PTSD may be more difficult than treating AUDs in the general population. The FDA-approved medication topiramate has been shown to improve drinking outcomes in people with AUDs. Topiramate has also improved symptoms in people with PTSD. This study is designed to investigate whether topiramate will improve drinking outcomes in Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Ages 21-64
* Diagnosis of PTSD via a score of 50 or higher on the Clinician Administered PTSD Scale (CAPS)
* Alcohol abuse or dependence per diagnosis in the medical record -or- by consuming more than 35 standard drinks per week over the previous 4 weeks as measured by the Timeline Follow-Back Interview
* A desire to reduce drinking behavior
* Any Race/Ethnicity

Exclusion Criteria:

* Currently taking a carbonic anhydrase inhibitor (e.g. zonisamide, acetazolamide, dichlorphenamide)
* Currently taking or have taken in the previous 3 months: acamprosate, naltrexone, disulfiram, topiramate
* Change in benzodiazepine dose within the previous 3 months
* Change in other (non-benzodiazepine) medication dose within the last 4 weeks
* Seizure disorder documented in the medical record
* Head trauma with loss of consciousness for greater than 30 minutes -or- a diagnosis of post-concussive syndrome documented in the medical record
* Suicide attempt within the previous 3 months or suicidal ideation within the previous 4 weeks
* A history of kidney stones
* A history of glaucoma
* ALT or AST liver enzymes elevated more than twice the upper limit of normal
* More than 4 unsuccessful attempts at inpatient alcohol treatment
* Medically unstable (including significant hypertension despite adequate treatment)
* A history of delirium tremens ("DTs") or alcohol withdrawal seizure
* Compulsory treatment to avoid legal consequences (e.g. imprisonment)
* Currently in a setting without access to alcohol (e.g. locked inpatient unit)

Ages: 21 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard A Fischer, M.D., Principal Investigator — Department of Veterans Affairs, University of Maryland School of Medicine
Locations (1):
- Baltimore VA, VA Maryland Health Care System, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants were withdrawn prior to assignment to a treatment group. Two did not return for study visits after signing consent and one did not meet eligibility criteria.
Period: Overall Study
Arm/Group | Topiramate | Placebo (Sugar Pill)
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo (Sugar Pill) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Heavy Drinking Days
Description: The Alcohol Timeline Follow Back (TLFB) interview was conducted to establish a baseline drinking pattern over the previous 90 days and confirm the presence of an alcohol use disorder (defined as consumption of greater than 35 standard drinks per week over the previous 4 weeks). The TLFB involves asking participants to retrospectively report their drinking days using a calendar.
Time Frame: 14 weeks
Population: There were not enough interested, eligible participants available to continue the study. Additionally, the study drug expired and the pharmacy that had done the compounding was bought by a larger chain and was set to be closed. Therefore, the study was stopped and closed in April 2013.
Arm/Group | Topiramate | Placebo (Sugar Pill)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Amount of PTSD Symptoms
Description: The Clinician Administered PTSD Scale (CAPS) contains 30 questions relating to PTSD symptoms. Each question asks about both the frequency and the severity of each symptom. These questions are split into categories. Each criterion has several questions, and scores for each criterion are added up at the end. To meet criteria for a symptom, a patient must meet criteria in both frequency and intensity score for each item. Frequency and intensity and then combined to form a single severity score. Severity scores range from 0-4, with 0 being absent to 4 being extreme/incapacitating.
Time Frame: 14 weeks
Population: as for outcome 1
Arm/Group | Topiramate | Placebo (Sugar Pill)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Topiramate | Placebo (Sugar Pill)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=1) | Placebo (Sugar Pill) (N=0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Subject evaluated by the PI and VA emergency department but was not admitted. Subject stopped taking study medication so determined not related to study drug or placebo.
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Severe nausea determined possibly related to study drug.
Dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Moderate dizziness determined to be possibly related to study drug.
Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Moderate stiffness determined to be possibly related to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No